CLINICAL TRIAL: NCT00003278
Title: Primary Central Nervous System Non-Hodgkins's Lymphoma (PCNSL): A Phase II Clinical Trial of Radiation Therapy and High Dose Corticosteroids for Elderly Patients (70 Years of Age and Older)
Brief Title: Radiation Therapy and High-Dose Corticosteroids in Treating Older Patients With Primary CNS Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-967351; CDR0000066184 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma; intraocular lymphoma
MeSH Terms: conditions — Lymphoma; Intraocular Lymphoma | interventions — Dexamethasone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiation + dexamethasone (Experimental): Patients undergo whole-brain radiotherapy (WBRT) daily 5 days a week for 4.5 weeks. Beginning 30 days after WBRT is completed, patients receive high-dose dexamethasone IV on days 1-5 during course 1 and on day 1 only during all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients are followed at 1 month after radiotherapy, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.
  Interventions: Drug: dexamethasone; Radiation: radiation therapy

INTERVENTIONS:
Drug: dexamethasone
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with a corticosteroid, such as dexamethasone, may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy and high-dose dexamethasone in treating older patients with primary CNS non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the effectiveness of high-dose dexamethasone after whole-brain radiotherapy in maintaining response and preventing recurrence in elderly patients with primary central nervous system non-Hodgkin's lymphoma.
* Assess the toxic effects of this regimen in these patients.
* Assess the survival rate of patients after this regimen.
* Identify the anatomic rates of recurrence and frequency of systemic involvement in patients treated with this regimen.
* Identify the factors that appear to be associated with outcome in patients treated with this regimen.

OUTLINE: Patients undergo whole-brain radiotherapy (WBRT) daily 5 days a week for 4.5 weeks. Beginning 30 days after WBRT is completed, patients receive high-dose dexamethasone IV on days 1-5 during course 1 and on day 1 only during all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month after radiotherapy, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed non-Hodgkin's lymphoma with intracranial lesions

  * Intraocular lymphoma eligible, if not sole site of disease
  * No occult systemic lymphoma
* Measurable or evaluable disease by CT scan or MRI
* No neoplastic meningitis or gross spinal cord involvement

PATIENT CHARACTERISTICS:

Age:

* 70 and over

Performance status:

* ECOG 0-3

Other:

* No prior history of lymphoma
* No other active malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* HIV negative
* No active peptic ulcer disease
* No uncontrolled diabetes mellitus
* No active pancreatitis
* No active bleeding
* No poorly controlled major psychiatric illness
* No serious uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow transplantation

Chemotherapy:

* No prior chemotherapy

Radiotherapy:

* No prior radiotherapy to the brain or head and neck region

Surgery:

* No prior transplantations (renal, hepatic, or cardiac)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 1998-03; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian P. O'Neill, MD, Study Chair — Mayo Clinic
Locations (14):
- United States (13):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - Medcenter One Health System, Bismarck, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] O'Neill BP, Habermann TM, Witzig TE, Rodriguez M. Prevention of recurrence and prolonged survival in primary central nervous system lymphoma (PCNSL) patients treated with adjuvant high-dose methylprednisolone. Med Oncol. 1999 Sep;16(3):211-5. doi: 10.1007/BF02906134. PMID 10523802
- [Result] Laack NN, Ballman KV, Brown PB, O'Neill BP; North Central Cancer Treatment Group. Whole-brain radiotherapy and high-dose methylprednisolone for elderly patients with primary central nervous system lymphoma: Results of North Central Cancer Treatment Group (NCCTG) 96-73-51. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1429-39. doi: 10.1016/j.ijrobp.2006.03.061. PMID 16863926
- [Result] Laack NN, Ballman KV, Brown PD, et al.: Toxicity of whole-brain radiotherapy (WBRT) and high-dose methylprednisolone (HDMP) for elderly patients (70 years of age and older) with primary central nervous system lymphoma (PCNSL): results of North Central Cancer Treatment Group (NCCTG) 967351. [Abstract] Neuro-Oncology 6 (4): RT-11, 361, 2004.